CLINICAL TRIAL: NCT03004586
Title: Endobronchial Ultrasound-guided Transbronchial Needle Aspiration Using a 22 vs 25-Gauge Needle; A Randomized Controlled Trial
Brief Title: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration Using a 22 vs 25-Gauge Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2016-0561; NCI-2017-00624 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Malignant Neoplasm of Respiratory and Intrathoracic Organ Carcinoma; Lung Cancer
Keywords: Malignant Neoplasm of Respiratory and Intrathoracic Organ Carcinoma; Lung cancer; Ultrasound-guided transbronchial needle aspiration; EBUS-TBNA; 25-gauge needle; 22-gauge needle
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS-TBNA:First Using a 25-Gauge Needle Then 22-gauge Needle (Experimental): Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed by first using a 25-gauge needle, followed by a 22-gauge needle.
  Interventions: Device: 25-Gauge Needle; Device: 22-Gauge Needle; Procedure: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration (EBUS-TBNA)
- EBUS-TBNA:First Using a 22-Gauge Needle Then 25-gauge Needle (Experimental): Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed by first using a 22-gauge needle, followed by a 25-gauge needle.
  Interventions: Device: 25-Gauge Needle; Device: 22-Gauge Needle; Procedure: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration (EBUS-TBNA)

INTERVENTIONS:
Device: 25-Gauge Needle — Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed by using a 25-gauge needle.
Device: 22-Gauge Needle — Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed by using a 25-gauge needle.
Procedure: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration (EBUS-TBNA) — Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) performed.
  Other Names: EBUS-TBNA

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of a smaller, 25-gauge needle when used in an endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) instead of a standard 22-gauge needle.

The safety of the needles will also be studied.

DETAILED DESCRIPTION:
As a part of participant's standard-of-care, participant will have a bronchoscopy of lesions on participant's lung nodules and/or lymph nodes before the EBUS-TBNA. Participant will sign a separate consent for the bronchoscopy.

If participant agrees to take part in this study, before participant's bronchoscopy, participant will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If participant is in Group 1, participant will have the EBUS-TBNA performed by first using a 25-gauge needle, followed by a 22-gauge needle.
* If participant is in Group 2, participant will have the EBUS-TBNA performed by first using a 22-gauge needle, followed by a 25-gauge needle.

To perform an EBUS-TBNA, a needle is inserted into the affected area using ultrasound imaging to collect tissue from the lungs and lymph nodes. The doctor will use the imaging to guide the needle into the area.

Length of Study:

Participation on the study will be over after the bronchoscopy and EBUS-TBNA.

This is an investigational study. The 22-gauge and 25-gauge needles are FDA approved for use in EBUS-TBNAs. The comparison of the 2 needles for this procedure is investigational. The study doctor can explain how the needles are designed to work.

Up to 120 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Indication for EBUS-guided needle biopsy based on suspicion of either benign or malignant disease in mediastinal or hilar lymph nodes.

Exclusion Criteria:

1. Patients who are pregnant or lactating
2. Inability to give informed consent
3. Patients in which only one lymph node station is expected to be sampled by the performing clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A. Eapen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 61 patients were enrolled with a total of 200 lymph node stations evaluated. We randomized the "needle size order" on a per-patient basis with first three needle passes performed with one needle and the remaining 4th and 5th needle passes performed with the other needle. All participants completed the studies and there were no dropouts. Since the randomization was done at the lymph node level, both arms had equal number of participants.
Units Other Than Participants: Lymph nodes
Groups:
- Intervention Group: First Using a 25-gauge Needle Then 22-gauge Needle: Participants in this group had their lymph nodes sampled with 25-gauge needle first followed by the 22-gauge needle.
- Control Group: First Using a 22-gauge Needle Then 25-gauge Needle: Participants in this group had their lymph nodes sampled with 22-gauge needle first followed by the 25-gauge needle.
Period: Overall Study
Arm/Group | Intervention Group: First Using a 25-gauge Needle Then 22-gauge Needle | Control Group: First Using a 22-gauge Needle Then 25-gauge Needle
Started | 31; 200 Lymph nodes | 30; 200 Lymph nodes
Completed | 31; 200 Lymph nodes | 30; 200 Lymph nodes
Not Completed | 0; 0 Lymph nodes | 0; 0 Lymph nodes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lymph nodes
Groups:
- All Study Participants: Participants had their lymph nodes sampled both with 25-gauge needle first followed by the 22-gauge needle and 22-gauge needle first followed by the 25-gauge needle.
Arm/Group | All Study Participants
Number analyzed (Participants) | 61
Number analyzed (Lymph nodes) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 61
Lymph Nodes Station [Number; unit: lymph nodes]
  Lymph Node Station: 11Rs | 21
  Lymph Node Station: 11Ri | 12
  Lymph Node Station: 10R | 1
  Lymph Node Station: 4R | 39
  Lymph Node Station: 2R | 7
  Lymph Node Station: 7 | 53
  Lymph Node Station: 4L | 27
  Lymph Node Station: 10L | 3
  Lymph Node Station: 11L | 35
  Lymph Node Station: 1 | 1
  Lymph Node Station: Mass (central) | 1
CT Scan Nodal Diameter Short Axis (mm) [Mean (Standard Deviation); unit: millimeters] | 9.1 (5.1)
EBUS Nodal Diameter Short Axis (mm) [Mean (Standard Deviation); unit: millimeters] | 9.5 (4.7)
Lymph Node Characteristic [Mean (Standard Deviation); unit: lymph nodes]
  Lymph Node Characteristic: Normal | 94 (47.0)
  Lymph Node Characteristic: Tumor (Cohesive) | 24 (12)
  Lymph Node Characteristic: Tumor (Dis-cohesive) | 11 (5.5)
  Lymph Node Characteristic: Granulomas/Sclerotic | 6 (3.0)
  Lymph Node Characteristic: Non-diagnostic | 10 (5.0)
Final Diagnosis [Number; unit: lymph nodes]
  Final Diagnosis: Inadequate/Non-diagnostic | 6
  Final Diagnosis: Normal Lymphoid Tissue | 128
  Final Diagnosis: Granulomatous Inflammation | 31
  Final Diagnosis: Necrosis | 1
  Final Diagnosis: Malignancy | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lymph Nodes With Adequate Samples
Description: The primary outcome was the proportion of concordance between the 22-gauge and 25-gauge needles in sample adequacy after two passes. The intervention group each of the lymph nodes sampled first with 25 gauge-needle, then the 22 gauge-needle. The Control Group each of the 200 lymph nodes were sampled first with the 22 gauge- needles, then the 25 gauge-needle. Sample adequacy was assessed after 2 passes using each needle in all participants and recorded.
Time Frame: One to two hours.
Population: All participants underwent sampling with both needles.
Measure: Number; unit: Percentage of Lymph Nodes
Units Other Than Participants: Lymph Nodes
Arm/Group | Intervention Group: First Using a 25-gauge Needle Then 22-gauge Needle | Control Group: First Using a 22-gauge Needle Then 25-gauge Needle
Number analyzed (Participants) | 31 | 30
Number analyzed (Lymph Nodes) | 200 | 200
Percentage of Lymph Nodes | 79 | 78.5

2. Secondary Outcome: Concordance With the Final Diagnosis
Description: The difference in the diagnostic yield between the 22-gauge and 25-gauge needles in terms of degree of concordance with the final diagnosis. The intervention group each of the lymph nodes sampled first with 25 gauge-needle, then the 22 gauge-needle. The Control Group each of the 200 lymph nodes were sampled first with the 22 gauge- needles, then the 25 gauge-needle. The percentage of concordance was calculated by comparing the 2 passes from each needle to the final diagnosis.
Time Frame: One to two hours
Population: All participants underwent sampling with both needles.
Measure: Number; unit: Percentage of concordance
Units Other Than Participants: Lymph Nodes
Arm/Group | Intervention Group: First Using a 25-gauge Needle Then 22-gauge Needle | Control Group: First Using a 22-gauge Needle Then 25-gauge Needle
Number analyzed (Participants) | 31 | 30
Number analyzed (Lymph Nodes) | 200 | 200
Percentage of concordance | 82 | 80.5

3. Secondary Outcome: Usability of the Needle
Description: The difference in usability between the 22-gauge and 25-gauge needles. All participant's lymph nodes were sampled by two 25-gauge needles and two 22-gauge needles for a total of 4 needles per person. Measured by a Likert scale 1-5 with 1 being the lowest and 5 being the maximum score. The intervention group each of the lymph nodes sampled first with 25 gauge-needle, then the 22 gauge-needle. The Control Group each of the 200 lymph nodes were sampled first with the 22 gauge- needles, then the 25 gauge-needle. The participants are reported per intervention.
Time Frame: 1-2 hours (Intra procedurally)
Population: Participant's lymph nodes were sampled by two 25-gauge needles and two 22-gauge needles for a total of 4 needles per person.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Needles
Groups:
- Intervention Group: First Using a 25-gauge Needle Then 22-gauge Needle: Participants lymph nodes were sampled first by two 25-gauge needles then two 22-gauge needles for a total of 4 needles per person.
- Control Group: First Using a 22-gauge Needle Then 25-gauge Needle: Participants lymph nodes were sampled first by two 22-gauge needles then two 25-gauge needles for a total of 4 needles per person.
Arm/Group | Intervention Group: First Using a 25-gauge Needle Then 22-gauge Needle | Control Group: First Using a 22-gauge Needle Then 25-gauge Needle
Number analyzed (Participants) | 61 | 61
Number analyzed (Needles) | 122 | 122
units on a scale
  Ease of needle insertion | 4.27 (0.85) | 4.95 (0.20)
  Visibility of the sheath | 4.58 (0.65) | 4.00 (0.81)
  Scope flexibility | 4.40 (0.87) | 4.65 (0.64)
  Ultrasound image quality | 4.62 (0.70) | 4.65 (0.65)
  Ease of needle puncture | 4.57 (0.75) | 4.53 (0.60)
  Ultrasound image quality following needle insertion | 4.62 (0.70) | 4.65 (0.65)
  Ease of needle removal | 4.71 (0.54) | 4.99 (0.11)

ADVERSE EVENTS:
Time Frame: within 24 hours of procedure
Description: adverse events were monitored for irrespective of specific needle intervention and therefore cannot be reported separately
Groups:
- Intervention Group: First Using a 25-gauge Needle Then 22 Gauge-needle: Participants lymph nodes sampled with 25-gauge needle first followed by the 22-gauge needle and sampled with 22-gauge needle first followed by the 25-gauge needle.
- Control Group: First Using a 22-gauge Needle Then 25 -Gauge Needle: Patients in this group had their lymph nodes sampled with 22-gauge needle first followed by the 25-gauge needle.
Arm/Group | Intervention Group: First Using a 25-gauge Needle Then 22 Gauge-needle | Control Group: First Using a 22-gauge Needle Then 25 -Gauge Needle
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03004586/Prot_SAP_000.pdf